CLINICAL TRIAL: NCT02506998
Title: Evaluation of Quality of Life in Allergic Rhinoconjunctivitis Patients Treated With Dialyzable Leukocyte Extracts as an Adjuvant
Brief Title: Quality of Life in Allergic Rhinoconjunctivitis Patients Treated With Dialyzable Leukocyte Extracts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Polytechnic Institute, Mexico (Other)
Collaborators: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Principal Investigator, Maria C Jimenez Martinez, MD PhD, National Polytechnic Institute, Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC-13-001
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergic rhinoconjunctivitis; Dialyzable Leukocyte Extracts
MeSH Terms: interventions — Transfer Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DLE plus standard medications (Experimental): DLE + Second generation anti histamines + Nasal corticosteroids DLE 2mg/5 milliliters (mL) P.O. every 24h per 5 days, followed by 2 mg/mL P.O. twice weekly for 5 weeks, follow by 2 mg/5mL per week for 5 weeks.
  Second generation anti histamines at standard dosis every 24h, and Nasal corticosteroids two spray released per nostril every 24 h per 11 weeks
  Interventions: Biological: DLE; Other: Second generation anti histamines + Nasal corticosteroids

INTERVENTIONS:
Biological: DLE — Adjuvant treatment
  Other Names: Transfer Factor; Transferon
Other: Second generation anti histamines + Nasal corticosteroids — Standard treatment

SUMMARY:
The purpose of this study is to determine the changes of quality of life of patients with allergic rhinoconjunctivitis treated with standard medications plus Dialyzable Leukocyte Extracts (DLE). All patients will receive DLE in combination with current guide lines-suggested standard medication.

DETAILED DESCRIPTION:
DLE are heterogenous mixtures of peptides under 10 kilo Daltons (kDa) obtained after disruption of peripheral blood leukocytes from healthy human donors. DLE have been reported to improve clinical response in allergies, such as asthma and atopic dermatitis.

The therapeutic effect of DLE is related to an immune modulatory effect that changes innate signaling pathways, such as Toll Like Receptors, and Nuclear Factor -kappa B; production of cytokines might also be modified with the use of DLE, including Tumor Necrosis Factor a, Interleukin (IL)-6, and induction of Interferon-g secretion, driving immune response to a T-helper Th1 immune-regulatory response, and thus helping to reduce allergy symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of symptomatic seasonal or perennial allergic rhinitis
* Active rhinoconjunctivitis
* Six week standard treatment before inclusion
* Confirmation of an Immunoglobulin E-mediated response through previous positive skin or in vitro allergen testing

Exclusion Criteria:

* Other immunological immune-mediated diseases such as autoimmune diseases and cancer.
* Unstable chronic disease, such as diabetes, cardiac diseases, chronic kidney failure, chronic hepatic disease.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 11 weeks
  Quality of Life evaluated by Standardized Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ(s)) Spanish version for Mexico

CONTACTS AND LOCATIONS:
Overall Officials: Toni Homberg, MD, Principal Investigator — National Polytechnic Institute

REFERENCES:
- [Derived] Homberg TA, Lara I, Andaluz C, Cervantes-Trujano E, Hernandez-Martinez PM, Perez-Tapia SM, Jimenez-Martinez MC. Quality of life in adult patients using dialyzable leukocyte extract for allergic rhinitis. Medicine (Baltimore). 2023 Jul 7;102(27):e34186. doi: 10.1097/MD.0000000000034186. PMID 37417619